CLINICAL TRIAL: NCT06984159
Title: An Open-Label, Single-Arm, Multicenter Clinical Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Leuprolide Injectable Emulsion in Advanced Prostate Cancer
Brief Title: The Study Will Evaluate if Leuprolide Mesylate is Safe and Effective in the Treatment of Subjects With Advanced Prostate Carcinoma, When Administered as Two Injections Six Months Apart.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GenSci093-6M
Record Dates: First submitted 2025-05-11; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Advanced Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Leuprolide Injectable Emulsion (Experimental)
  Interventions: Drug: Leuprolide Injectable Emulsion (CAMCEVI®)

INTERVENTIONS:
Drug: Leuprolide Injectable Emulsion (CAMCEVI®) — Leuprolide Injectable Emulsion (CAMCEVI®)，Subcutaneous injection，Once every 24 weeks for a total of 2 doses

SUMMARY:
Evaluate the Safety, Efficacy and Pharmacokinetics of Leuprolide Injectable Emulsion in Advanced Prostate Cancer

ELIGIBILITY:
Inclusion Criteria:

* After having the scope and nature of the study explained, subjects must voluntarily sign the ICF prior to the screening visit and be willing to comply with the study requirements and cooperate with all scheduled tests
* Male, aged ≥ 18 years old.
* Pathologically confirmed advanced prostate cancer candidate for Androgen Deprivation Therapy, including patients those who have undergone radical treatment (surgical resection, external radiotherapy, or cryotherapy).

Exclusion Criteria:

* Received or are undergoing Androgen Deprivation Therapy (surgical castration or drug Androgen Deprivation Therapy including but not limited to gonadotropin-releasing hormone [GnRH] receptor agonists, GnRH receptor antagonists, estrogen and progesterone and their analogs, androgen receptor antagonists, androgen synthesis inhibitors, etc.).
* Major surgery (including but not limited to radical prostatectomy, etc.), radiotherapy, chemotherapy, immunotherapy, cryotherapy, etc. within 4 weeks prior to the screening visit, or plan to receive the above treatments during the study
* Receipt of any vaccination within 4 weeks prior to first dose (except COVID-19 vaccination).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Cumulative probability of maintaining serum testosterone at a castrate level (≤ 50 ng/dL) from the end of 28 days after the first dose to the end of 168 days after the second dose. | from the end of 28 days after the first dose to the end of 168 days after the second dose.
  To evaluate the castrate level maintenance of Leuprolide Injectable Emulsion from the end of 28 days after the first dose to the end of 168 days after the second dose, with serum testosterone as a surrogate parameter for the assessment of efficacy and a castrate level of 50 ng/dL.
including but not limited to:adverse events (AEs) and serious adverse events (SAEs), vital signs, physical examination, laboratory tests, 12-lead electrocardiogram (ECG), injection site reactions, local tolerance, etc. | 336 days
  To evaluate the safety and tolerability of Leuprolide Injectable Emulsion after two subcutaneous injections in patients with advanced prostate cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China